CLINICAL TRIAL: NCT04708262
Title: A Case-Series Examination of a Brief CAT-Informed Intervention (CATCH-Y) for Young People That Have Self-Injured
Acronym: CATCHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Peter Taylor, Dr, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 287611
Record Dates: First submitted 2021-01-06; First posted 2021-01-13 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Non-Suicidal Self Injury
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Single group case series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Analytic Therapy for Containing Self-Harm in Young People (Experimental): Brief one-to-one psychological therapy using Cognitive Analytic Therapy principles, designed for young people who self-harm
  Interventions: Other: Cognitive Analytic Therapy for Containing Self-Harm in Young People

INTERVENTIONS:
Other: Cognitive Analytic Therapy for Containing Self-Harm in Young People — The intervention will run over five sessions, each lasting around 30 - 40 minutes. Researchers will follow the CATCH-Y manualised treatment guide. CATCH-Y is a brief, five session psychological intervention based upon CAT principles and designed to help young people who have self-injured.

SUMMARY:
Non-suicidal self-injury (NSSI), the term used for when somebody purposefully hurts themselves without intending to end their life. Often, it suggests that there are other difficulties going on in someone's life. Talking therapies can be offered to help however currently there is little evidence to show which therapies help most. CATCH-Y (Cognitive Analytic Therapy for Containing Self-Harm in Young People) is a brief talking therapy which has been created to support young people who self-injure. It aims to help young people and those around them build to a shared understanding of their difficulties. Previously a group of adults, who have a history of self-harm, have engaged in a trial version of CATCH-Y for adults, in which it was found to be positive, safe and feasible.

The study will aim to recruit nine young people who have self-injured in the past. Participants must be aged between 13 - 17 years old and have self-injured within the last six months. They will be recruited from local Child and Adolescent Mental Health Services (CAMHS) and associated 3rd sector organisations. The therapy is five sessions long, with two assessment sessions before the therapy begins and one assessment session post-therapy. Online assessments will be completed throughout. CATCH-Y involves working with the therapist to understand a young person's past and current experiences, linked to their self-injurious behaviours. This individualised approach could benefit these young people.

As a novel treatment, and in accordance with the medical research council (MRC) framework, the feasibility and acceptability of CATCH-Y should be considered before progressing to a larger trial. This trial will examine the feasibility and acceptability of the CATCH-Y intervention through attendance and retention rates, data completion and intervention acceptability. As a secondary measure, the trial will investigate whether CATCH-Y shows preliminary evidence for positive change.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be between the ages of 13 - 17 years.
* Participants will have self-injured at least once in the past six months and have a lifetime history of two or more episodes of NSSI.
* Participants will have a clinician allocated to them within CAMHS or a 3rd sector service.
* Participants will have access to the Internet.

Exclusion Criteria:

* Participants will be excluded if they are currently receiving alternative psychological therapies from a mental health professional. Participants may be receiving other forms of ongoing contact and support that do not constitute a formal psychological therapy.
* Participants will be excluded if they have a severe intellectual disability, which would impair their ability to participate without considerable adaptations being made to the intervention.
* Participants will be excluded if they have inadequate English-language speaking skills due to limitations in their ability to engage with talking therapies in the English language.
* Participants will be excluded if they are judged at high risk of harm to themselves, operationalised as having current suicidal thoughts with a high intent or active plan to end their life.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Retention rate | seven weeks
  Attendance at each session will be recorded to determine whether over 70 percent of participants will be retained from baseline to the end of the study.
Referral rates | Completion of study, approximately 18 months
  Referrals will be recorded to test the hypothesis that over 50 percent of those who are referred to the study and are eligible to participate, consent to take part.
Missing data | Completion of study, approximately 18 months
  Completion of measurements will be analysed to test whether the level of missing data exceeds 20 percent per assessment.
Acceptability | up to 12 weeks
  An exploration of factors that influence engagement (including what was helpful/unhelpful) will be determined in the adapted version of the client satisfaction questionnaire. Response frequencies, and qualitative comments, will be presented item by item.

SECONDARY OUTCOMES:
Repertory Grid | up to 12 weeks
  Repertory grids: The repertory grid will be used to explore changes in participants' perceptions of the self, others and their experiences of NSSI. Participants will be asked to complete them prior to, and following, completion of CATCH-Y. This assessment will be completed as a structured interview, with one of the researchers talking through and explaining each step. The repertory grids will be developed following established techniques (Jankowicz, 2003). Previously repertory grids have been used with adolescents (Sewell, 2020). These measures will be used pre and post intervention.
Motivation for Youth Treatment Scale | up to 12 weeks
  Motivation for Youth Treatment Scale. This evaluates motivation to change and desire to find solutions to difficulties in youths and their caregivers. A psychometric evaluation of this scale conducted with young people aged 11-18 found it to be a reliable tool for assessing important dimensions of intrinsic treatment motivation (Breda & Riemer, 2012). This measure will be assessed online using select survey, pre and post intervention. The minimum score is 1, the maximum score is 40. Higher scores mean a better outcome (improved motivation).
Recovery Questionnaire | up to 12 weeks
  Recovery Questionnaire. Examines recovery of functionality and outlook post-treatment. An evaluation of the psychometric properties of the Recovery Questionnaire with 65 young people showed good internal consistency and test-retest reliability (Bentley, Bucci & Hartley, 2019). This measure will be assessed online using select survey, pre and post intervention. The minimum score is 0, the maximum score is 93. Higher scores mean a better outcome (improved recovery).
Alexian Brothers Urges to Self-injure scale (ABUSI) | up to 12 weeks
  Alexian Brothers Urges to Self-injure scale (ABUSI): A measure to assess the frequency, intensity and duration of the urge to self-injure. The ABUSI has shown good internal consistency and reliability (Chavez-Flores et al., 2019). In addition, a recent study found that the ABUSI provided valid information in a population of students who self-injured (Dimitrova, Radkova, Stoyanov & Petrov, 2020). This measure will be assessed online using select survey, pre, post and weekly during the intervention. It will also be assessed for four weeks post-intervention. Summed scores range from 0 to 30 with higher scores indicating greater urges (poorer outcome).
Patient Health Questionnaire for Adolescents (PHQ-9A) | up to 12 weeks
  Patient Health Questionnaire for Adolescents (PHQ-9A): Low mood clinical evaluation. An examination of the PHQ-9A completed by 442 young people, showed positive validity of the measure (Richardson et al., 2010). This measure will be assessed online using select survey, pre, post and weekly during the intervention. It will also be assessed for four weeks post-intervention. Summed scores range from 0 to 27 with higher scores indicating lower mood (poorer outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Given small scale of the study there are no plans to make the data available to other researchers